CLINICAL TRIAL: NCT07343492
Title: Individualized fMRI and Molecular Profiling Reveal Functional Preservation in Glioma Peritumoral Edema
Brief Title: fMRI Reveal Functional Preservation in Glioma Peritumoral Edema
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Simin Zhang, prof, West China Hospital
Other Study IDs: 82271961
Record Dates: First submitted 2025-12-20; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diffuse Glioma Patients

SUMMARY:
he goal of this observational study is to investigate the functional and biological characteristics of the brain tissue surrounding diffuse gliomas, known as peritumoral edema (PTE). The study aims to determine if a non-invasive brain imaging technique, resting-state functional MRI (rs-fMRI), can identify which parts of this edematous tissue are functionally preserved. The main questions it aims to answer are:

Can individualized rs-fMRI mapping accurately distinguish functionally active subregions from non-functional subregions within the peritumoral edema?

Do these functionally preserved regions, identified by imaging, correspond to areas with lower tumor cell infiltration and higher neuronal integrity when examined microscopically?

Participants prospectively enrolled for glioma resection surgery as part of their standard clinical care will undergo preoperative rs-fMRI. This imaging data will be used to create individualized functional network maps of the PTE. During the planned surgery, biopsies will be taken from PTE areas identified by the rs-fMRI analysis as "functionally preserved" and "non-preserved." These tissue samples will then undergo molecular analysis to assess markers for tumor proliferation (Ki-67), invasiveness (Nestin), neuronal integrity (NeuN), and synaptic density (PSD-95, Synapsin-1). Finally, the functional characteristics derived from the preoperative imaging will be correlated with the molecular profiles of the corresponding tissue samples.

ELIGIBILITY:
Inclusion Criteria:

Right-handedness Pathologically confirmed diffuse glioma (WHO grade 2-4, based on 2021 WHO classification) Clinical indication for preoperative MRI Clearly delineated FLAIR hyperintensity surrounding the tumor Age 18 years or older Willing and able to provide written informed consent

Exclusion Criteria:

Prior brain biopsy or treatment for glioma Contraindications to MRI (e.g., pacemaker, ferromagnetic implants, severe claustrophobia) Comorbid psychiatric or neurological conditions that may affect functional imaging Head motion exceeding 1.0 mm translation or 1.0° rotation during rs-fMRI acquisition Framewise displacement (FD) greater than 0.2 mm during rs-fMRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gliomas
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Functional connectivity strength of peritumoral edema regions measured by resting-state fMRI | 1-2 weeks before surgery
  Nodal connectivity strength between peritumoral edema (PTE) subregions and 17 canonical Yeo functional networks, computed from resting-state fMRI data using individualized functional parcellation. Connectivity strength is calculated as the Pearson correlation coefficient between mean BOLD time series.
Shannon entropy of edge-centric functional connectivity in peritumoral edema regions | 1-2 weeks before surgery
  Normalized Shannon entropy (range 0-1) calculated from edge-centric functional connectivity analysis, reflecting the diversity of edge community participation for peritumoral edema subregions. Higher entropy indicates greater integrative complexity.
Ki-67 proliferation index in functionally preserved versus non-preserved peritumoral edema regions | During surgery (intraoperative sampling)
  Percentage of Ki-67 positive cells assessed by immunofluorescence staining in intraoperative tissue samples from functionally preserved and non-functionally preserved PTE compartments.
Synaptic marker expression (PSD-95, Synapsin-1) in peritumoral edema subregions | During surgery (intraoperative sampling)
  Percentage of PSD-95 and Synapsin-1 positive cells assessed by immunofluorescence in paired tissue samples from functionally preserved and non-preserved PTE regions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided